CLINICAL TRIAL: NCT03065088
Title: The PreventIT Feasibility Randomised Controlled Trial in Young Older Adults, Comparing Two Lifestyle-integrated Exercise Interventions Delivered by Use of ICT or an Instructor, With a Control Group
Brief Title: The PreventIT Trial in Young Older Adults, Comparing Two Lifestyle-integrated Exercise Interventions
Acronym: PreventIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: VU University of Amsterdam (Other); Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); University of Bologna (Other); University of Manchester (Other); Local Centre Health Unit Tuscany (Unknown); Ecole Polytechnique Fédérale de Lausanne (Other); Doxee S.p.A. (Unknown); Health Leads BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016/1891
Record Dates: First submitted 2017-02-14; First posted 2017-02-27 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Young Older Adults
Keywords: Exercise; Feasibility Studies; Healthy Lifestyle; Health Promotion; Health Behavior; Aging; Activities of Daily Living; Mobile Applications
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: This is a feasibility study run as a randomised controlled trial (RCT). This is a multi-centre trial with three centres, Trondheim, Amsterdam, and Stuttgart, with two behaviour change exercise programmes (aLiFE and eLiFE) and a control group, with a 6 months intervention period and 6 month follow up.
Who Masked: Outcomes Assessor
Masking Description: Assessors are blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aLiFE (Experimental): The aLiFE programme is developed for young older adults, where balance activities, strengthening activities, and specific recommendations for increasing physical activity, are embedded within everyday activities, so that the activities can be performed multiple times throughout the day. The programme is presented by an instructor by use of a paper based manual during a 6 month intervention period in participants homes.
  Interventions: Behavioral: aLIFE
- eLiFE (Experimental): The aLiFE programme is transferred to a mobile health system, called the eLiFE. The intervention is delivered on smartphones and smartwatches including inertial sensors well suited to monitor physical activity and movement quality in daily life. An instructor teaches the participants how to use the mobile health system during home visits and phone calls during the 6 month intervention period. A virtual instructor teaches the participants the eLiFE programme. Pictures and videos of the aLiFE activities are delivered by use of the system. Behavioural change strategies are also included in the system.
  Interventions: Behavioral: eLIFE
- control (Active Comparator): The control group follows the World Health Organization's recommendations of physical activity.
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: aLIFE — The aLiFE programme is taught by an instructor during six home visits and 3 phone calls during the 6-month intervention period. The programme will be personalised by use of an initial balance and strength assessment (aLiFE assessment tool). The participants assigns activities to his or her daily activities, and during subsequent home visits, the number of activities and task demands are upgraded. Participants will be taught how to select opportunities themselves to embed activities into their individual daily routine, and how to progress over time.
  Arms: aLiFE
Behavioral: eLIFE — The eLIFE includes a personalised ICT-administered training schedule using the activities developed in aLiFE, delivered in the form of video clips, pictures and text/verbal instructions on a smartphone and smartwatch application. Personalisation of activity content will be decided based on a phenotype tool and initial difficulty level is decided through the aLiFE assessment tool. In addition, a virtual instructor teaches the participants how to carry out the eLiFE programme. The user receives motivational messages and feedback, and there will be a possibility for social interaction between the participants. The instructors teach the eLiFE participants the programme during 4 home visits and 3 phone calls during the 6 month intervention period.
  Arms: eLiFE
Behavioral: control — The control group follows the World Health Organization's recommendations of physical activity. The control participants will receive one home visit and be given a written letter with the activity recommendations.
  Arms: control

SUMMARY:
The feasibility randomised controlled trial is part of the EU funded project "PreventIT" (2016-2018) responding to the Horizon 2020, Personalised health and care (PHC), call PHC-21: Advancing active and healthy ageing with ICT: Early risk detection and intervention. The PreventIT project focuses on a new behaviour change activity approach for young older adults (61-70 years of age) with an overall aim of early prevention of functional decline and to empower people to take care of their own health.

DETAILED DESCRIPTION:
In this feasibility randomised controlled trial two interventions are compared with a control group. The aLiFE programme includes instructor and paper manual delivery of life-style integrated activities, while the eLiFE programme delivers the same activities by use of smartphone and smartwatch applications. The control group is asked to follow the World Health Organisation's physical activity recommendations.

The main aim is to assess feasibility of the aLiFE and eLiFE programmes and a second aim to suggest sample size and design for a future Phase III clinical trial.

OBJECTIVES: How is the feasibility of having young older adults (between 61-70 years) to perform the aLiFE and eLiFE interventions.

Specifically:

1. Participation: How is the adherence of specific activities and to the entire aLiFE and eLiFE interventions of young older adults?
2. Technology: How is the feasibility and usability of the eLiFE intervention delivered using smartphones and smartwatches as platform, regarding user interface, goal setting, feedback, motivational messages, and social interaction?
3. Outcome measures: How is the risk reduction of functional decline, measured by the Later Life Function and Disability Instrument and behavioural complexity, for the aLiFE and the eLiFE interventions compared to a control group, and what are the estimates of effect sizes for the primary and secondary study outcome measure?
4. Health economics evaluation: Is it feasible to collect data on, and estimate, health care resource utilization, costs and quality-adjusted life years (QALYs), and model incremental cost-effectiveness ratios (ICERs) of aLiFE, eLiFE compared with the control group over a 6-month, 12-month, and 24-month time horizon?

The study is approved by the three ethical sites prior to study start.

(October 3rd, 2017) The final Data Analysis Plan has been closed before the start of the first post-test assessment in the PreventIT feasibility RCT, starting on the 4th of October 2017.

ELIGIBILITY:
Inclusion Criteria:

* born in the years 1947-1956
* Retired (more than 6 months, <50% paid/unpaid work)
* Home-dwelling
* Able to read newspaper or text on smartphone
* Speak Norwegian/Dutch/German
* Able to walk 500 m without walking aids
* Available for home visits the following 6 weeks
* Defined "at risk" for functional decline by the risk screening instrument developed in the PreventIT project

Exclusion Criteria:

* Current participation in an organised exercise class >1 per week or moderate-intensity physical activity ≥150 min/week in the previous 3 months
* Travels planned >2mths during follow-up
* Cognitive impairment (MOCA <24 points)
* Medical conditions:

  1. Heart failure New York Heart Function Assessment (NYHA) class III and IV
  2. Acute myocardial infarction last 6 months or unstable angina
  3. Pericarditis, myocarditis, endocarditis in the last 6 months
  4. Symptomatic aortic stenosis
  5. Cardiomyopathy
  6. Resting blood pressures of a systolic >180 or diastolic >100 or higher
  7. Chronic Obstructive Pulmonary Disease (COPD) Gold class III and IV
  8. Uncontrolled Asthma (at least 2 exacerbation in the last 6 months)
  9. Amputated lower extremities
  10. On active cancer treatment during last 6 months
  11. Ankylosing spondylitis
  12. History of schizophrenia
  13. Parkinsons disease
  14. Recently diagnosed Cerebrovascular Accident (<6 months)
  15. Epilepsy (treated with medication)
  16. Severe rheumatic arthritis interfering with mobility
  17. Fracture of lumbar spine / thoracic spine or lower extremity in the last 6 months
  18. 3 fractures in the last 2 years due to severe osteoporosis

Ages: 61 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Self-reported function and disability | Change; baseline, 6 months and 12 months
  Measured using the Late-Life Function and Disability Instrument (LLFDI)
Behavioural complexity metric | Change; baseline, 6 months and 12 months
  A composite measure of physical activity, sleep, and social participation, measured by a unitless scale. Physical activity and sleep is objectively measured by activity monitors worn at the lower back and the wrist, while social interaction is assessed as phone calls.

SECONDARY OUTCOMES:
Balance and mobility | Change; baseline, 6 months and 12 months
  Assessed by the Community Balance and Mobility Scale (CB&M)
Static balance | Change; baseline, 6 months and 12 months
  Assessed by the Eight Level Balance Scale
Gait speed | Change; baseline, 6 months and 12 months
  will be measured during a 4 m walk at usual pace and 7m walk at usual and fast pace
Grip Strength | Change; baseline, 6 months and 12 months
  will be measured by the JAMAR dynamometer (kg)
Functional Leg Strength | Change; baseline, 6 months and 12 months
  assessed by the 5-chair stand
Cognitive function | Change; baseline, 6 months and 12 months
  assessed by the Montreal Cognitive Assessment Tool (MoCA)
Mood | Change; baseline, 6 months and 12 months
  Self-reported by use of the Center for Epidemiologic Studies Depression Scale (CES-D)
Fear of falling | Change; baseline, 6 months and 12 months
  short Falls Efficacy Scale-International (short FESI)
Health related quality of life | Change; baseline, 6 months and 12 months
  as assessed by the EuroQol - EQ-5D-5L
Health related quality of life | Change; baseline, 6 months and 12 months
  as assessed by the Short Form Quality of Life (SF-12)
Instrumented functional strength | Change; baseline, 6 months and 12 months
  Instrumented 30sec chair stand
Instrumented standing balance | Change; baseline, 6 months and 12 months
  Instrumented Static balance
Instrumented mobility | Change; baseline, 6 months and 12 months
  Instrumented Time up and go test (iTUG)
Number of participants completing the different parts of the study | Screening, baseline, 6 months, and 12 months follow up
  Flow of participants during the study (number of completers and drop outs at different phases of the study)
Adverse Events | Through study completion, an average of 12 months
  Numbers, description, and severity reported by the assessors and instructors
Experience with the interventions, including motivation and behaviour change | Baseline, 6 months, and 12 month follow up
  7-point Likert Scale
Experience with the interventions, including motivation and behaviour change | Baseline, 6 months, and 12 month follow up
  Focus group interview
Process evaluation | 12 months
  Focus group interview
Technology evaluation | 6 months and 12 month follow up
  the System Usability Scale
Technology evaluation | 6 months and 12 month follow up
  the Telehealthcare Satisfaction Questionnaire
Attendance and adherence intervention | From date of first home visit until the date of the 12 month follow-up, assessed up to 12 months
  Single question every four week (email or mail)
Quality Adjusted Life Years (QALYs) | Baseline, 6 months, and 12 month follow up
  Short Form Quality of Life (SF-12)
Quality Adjusted Life Years (QALYs) | Baseline, 6 months, and 12 month follow up
  EuroQol - EQ-5D-5L
Cost-effectiveness | Baseline, 6 months, and 12 month follow up
  Incremental cost-effectiveness ratios (ICERs)
Acceptance of self-administered tests | Baseline and 12 month follow up
  Self-assessment test battery for physical function
Accelerometer Collected percentages of sedentary time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected duration of sedentary time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected intensity (metabolic equivalent) of sedentary time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected percentages of walking time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected duration of walking time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected intensity (metabolic equivalent) of walking time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected percentages of active time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected duration of active time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors
Accelerometer Collected intensity (metabolic equivalent) of active time during 7 days | Change; baseline, 6 months and 12 months
  Objectively measured by activity monitors

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Helbostad, phd prof, Study Director — Norwegian Universitiy of Science and Technology
Locations (3):
- Klinik für Geriatrische Rehabilitation, Stuttgart, Germany
- MOVE Research Institute Amsterdam, Amsterdam Center on Aging, Amsterdam, Netherlands
- NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taraldsen K, Mikolaizak AS, Maier AB, Boulton E, Aminian K, van Ancum J, Bandinelli S, Becker C, Bergquist R, Chiari L, Clemson L, French DP, Gannon B, Hawley-Hague H, Jonkman NH, Mellone S, Paraschiv-Ionescu A, Pijnappels M, Schwenk M, Todd C, Yang FB, Zacchi A, Helbostad JL, Vereijken B. Protocol for the PreventIT feasibility randomised controlled trial of a lifestyle-integrated exercise intervention in young older adults. BMJ Open. 2019 Mar 20;9(3):e023526. doi: 10.1136/bmjopen-2018-023526. PMID 30898801
- [Derived] Mikolaizak AS, Taraldsen K, Boulton E, Gordt K, Maier AB, Mellone S, Hawley-Hague H, Aminian K, Chiari L, Paraschiv-Ionescu A, Pijnappels M, Todd C, Vereijken B, Helbostad JL, Becker C. Impact of adherence to a lifestyle-integrated programme on physical function and behavioural complexity in young older adults at risk of functional decline: a multicentre RCT secondary analysis. BMJ Open. 2022 Oct 5;12(10):e054229. doi: 10.1136/bmjopen-2021-054229. PMID 36198449
- [Derived] Taraldsen K, Mikolaizak AS, Maier AB, Mellone S, Boulton E, Aminian K, Becker C, Chiari L, Follestad T, Gannon B, Paraschiv-Ionescu A, Pijnappels M, Saltvedt I, Schwenk M, Todd C, Yang FB, Zacchi A, van Ancum J, Vereijken B, Helbostad JL. Digital Technology to Deliver a Lifestyle-Integrated Exercise Intervention in Young Seniors-The PreventIT Feasibility Randomized Controlled Trial. Front Digit Health. 2020 Jul 31;2:10. doi: 10.3389/fdgth.2020.00010. eCollection 2020. PMID 34713023
- [Derived] Gordt K, Nerz C, Mikolaizak AS, Taraldsen K, Pijnappels M, Helbostad JL, Vereijken B, Becker C, Schwenk M. Sensitivity to Change and Responsiveness of the Original and the Shortened Version of the Community Balance and Mobility Scale for Young Seniors. Arch Phys Med Rehabil. 2021 Nov;102(11):2102-2108. doi: 10.1016/j.apmr.2021.03.036. Epub 2021 Apr 29. PMID 33932360